CLINICAL TRIAL: NCT05898126
Title: Effect of Personalized Hemodynamic Management Based on Serum Renin Concentration on Acute Kidney Injury Progression in Patients With Shock: a Randomized Controlled Trial.
Brief Title: Renin-guided Hemodynamic Management in Patients With Shock
Acronym: RENIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Full Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RENIN - 141/INT/2022; GR-2021-12375069 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Shock
Keywords: Shock; Renin; Vasopressor; Lactate; Acute Kidney Injury; Intensive Care Unit; Mortality; Quality of life
MeSH Terms: conditions — Shock; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Clinical trial in which patients affected by shock, randomly receive either renin-guided hemodynamic management or usual care.
Who Masked: Participant
Masking Description: Single blind trial. Participants will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renin-guided hemodynamic management (Experimental): We will measure serum renin values every six hours. If the measured renin concentration increases by more that 20% compared with the last value, the target mean arterial pressure (MAP) will be elevated to 75-80 mmHg. If the subsequent renin level is still rising, the target MAP will be further raised to 85-90 mmHg and the addition of inotropes will be considered. If the first subsequent renin level decreases or increases by ≤20%, the target MAP will be kept at 75-80 mmHg. If the renin level at the subsequent measurement after reaching the highest step of management protocol is still increasing, a failure of the intervention will be declared, the target MAP will return to 65-70 mmHg. If renin level further decreases or increases ≤20% for two consecutive measurements, we will downgrade the target MAP to the previous step.
  Interventions: Procedure: Renin-guided hemodynamic management
- Usual care (Sham Comparator): Patients in the usual care group will be managed according to standard of practice at each participating center.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Renin-guided hemodynamic management — If normalization of renin levels is achieved (values within the normal laboratory range), we will continue with usual care according to local protocols.
  Arms: Renin-guided hemodynamic management
Procedure: Usual care — Standard of care
  Arms: Usual care

SUMMARY:
Shock is a major risk factor for mortality among patients admitted to intensive care units (ICUs). Since various hemodynamic strategies uniformly delivered to patients with shock have failed to improve clinically relevant outcomes, individualized approaches for shock supported by robust evidence are required. This study will be a prospective, multicenter, parallel-group, single-blind, randomized controlled trial. The investigators will randomly assign 800 critically ill patients requiring norepinephrine infusion to the renin-guided or usual care groups. The investigators hypothesize that renin-guided hemodynamic management, compared to usual care, can reduce a composite of mortality and acute kidney injury (AKI) progression in patients requiring vasopressor support.

DETAILED DESCRIPTION:
Shock is a common cause of death among patients admitted to intensive care units. Acute kidney injury (AKI) frequently occurs in patients with shock (3, 4). Maintaining adequate perfusion pressure and oxygen delivery is crucial in the hemodynamic management of shock (5). Several randomized controlled trials have evaluated the effect of various hemodynamic protocols treating shock patients with a "one size fits all" approach. However, such protocols did not reduce mortality (6-8). The task force of the surviving sepsis campaign identified the personalization of sepsis resuscitation as a research priority (9). Moreover, a large RCT showed that personalizing blood pressure targets reduced the risk of postoperative organ dysfunction in patients undergoing major surgery (10). These findings suggest that applying individualized hemodynamic strategy may optimize shock treatment and potentially improve outcomes (11).

Recent studies have investigated renin as a novel marker of tissue hypoperfusion in critically ill patients. While serum lactate level has been the most common and validated marker for tissue hypoperfusion (12), several studies are now suggesting that renin may predict mortality better than lactate in critically ill patients (13, 14). Notably, relative renin increase is associated with adverse clinical outcomes and shock reversal has been shown to decrease renin concentration (15).

The investigators aim to perform the Randomized Evaluation of persoNalized hemodynamIc maNagement based on serum renin concentration (RENIN) trial to test the hypothesis that renin-guided hemodynamic management can reduce a composite of mortality and acute kidney injury (AKI) progression during the hospital stay in patients requiring vasopressors compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Admitted to an intensive care unit (ICU)
* Requiring norepinephrine infusion at any dose to maintain a mean arterial pressure (MAP) of ≥65 mmHg after initial fluid resuscitation
* Expected to stay in the ICU for at least 24 hours
* Written informed consent from the patient him-/herself or the patient's next of kin as requested by the ethics committee.

Exclusion Criteria:

* Pregnancy
* Refused informed consent
* Current enrollment into another randomized controlled trial that does not allow concomitant enrollment
* Requiring vasopressors for >12 hours before the enrollment
* Renal failure with an imminent need for renal replacement therapy (RRT)
* Intention to use RRT by clinical judgment despite lack of urgent clinical indication
* AKI stage 2 and 3 at enrollment according to the KDIGO criteria
* Prior enrollment in this study
* Severe liver disease (Child-Pugh score >7 points)
* Chronic kidney disease (CKD) equal to or worse than CKD stage IV (eGFR <30 mL/min/1.73 m2)
* History of kidney transplant
* Any condition explicitly requiring a higher or lower blood pressure target according to clinical judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2027-07-28 (Estimated)

PRIMARY OUTCOMES:
A composite of mortality or AKI progression at 30 days after randomization. | 30 days
  The primary outcome will be a composite of mortality or AKI progression at 30 days after randomization. We will define AKI progression as increasing at least two AKI stages compared to the AKI stage at study enrollment. We will define and stage AKI according to the current international criteria, the KDIGO guidelines (16). We will use both creatinine and urine output criteria.

SECONDARY OUTCOMES:
All-cause mortality at intensive care unit discharge, hospital discharge, and 90 days after randomization. | 90 days
The need for and duration of vasopressors at 30 days after randomization | 30 days
  Deaths within the initial 30 days were assigned 30 days of duration of vasopressors at day 30.
Days alive and free from mechanical ventilation | 30 days
  Deaths within the initial 30 days were assigned zero days alive and free from mechanical ventilation at day 30.
Day alive and free from renal replacement therapy. | 30 days
  Deaths within the initial 30 days were assigned zero days alive and free from renal replacement therapy at day 30.
Days alive and outside the ICU. | 30 days
  Deaths within the initial 30 days were assigned zero days alive and outside the ICU at day 30.
Duration of hospital stay. | 30 days
  Deaths within the initial 30 days were assigned 30 days of hospital stay.
Major adverse kidney events at day 90. | 90 days
  Major adverse kidney events are defined as a composite of death, the dependence of renal replacement therapy, and persistent renal dysfunction (defined as a 25% or greater decline in estimated glomerular filtration rate (eGFR) from the baseline) (17).
Quality of life at day 90. | 90 days
  EQ-5D-5L is the most widely used measure of health-related quality of life.
Adverse events during hospital stay. | 30 days
  Adverse events will include atrial fibrillation, acute myocardial infarction, ventricular fibrillation or tachycardia, digital ischemia, mesenteric ischemia, bleeding, reintubation, need for non-invasive ventilation, delirium, and stroke.

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospital Dubrava, Dubrava, Croatia
- Italy (2):
  - Ospedale Mater Domini, Catanzaro, Calabria
  - IRCCS Ospedale San Raffaele, Milan

REFERENCES:
- [Background] Orban JC, Walrave Y, Mongardon N, Allaouchiche B, Argaud L, Aubrun F, Barjon G, Constantin JM, Dhonneur G, Durand-Gasselin J, Dupont H, Genestal M, Goguey C, Goutorbe P, Guidet B, Hyvernat H, Jaber S, Lefrant JY, Malledant Y, Morel J, Ouattara A, Pichon N, Guerin Robardey AM, Sirodot M, Theissen A, Wiramus S, Zieleskiewicz L, Leone M, Ichai C; AzuRea Network. Causes and Characteristics of Death in Intensive Care Units: A Prospective Multicenter Study. Anesthesiology. 2017 May;126(5):882-889. doi: 10.1097/ALN.0000000000001612. PMID 28296682
- [Background] Mayr VD, Dunser MW, Greil V, Jochberger S, Luckner G, Ulmer H, Friesenecker BE, Takala J, Hasibeder WR. Causes of death and determinants of outcome in critically ill patients. Crit Care. 2006;10(6):R154. doi: 10.1186/cc5086. PMID 17083735
- [Background] Marenzi G, Assanelli E, Campodonico J, De Metrio M, Lauri G, Marana I, Moltrasio M, Rubino M, Veglia F, Montorsi P, Bartorelli AL. Acute kidney injury in ST-segment elevation acute myocardial infarction complicated by cardiogenic shock at admission. Crit Care Med. 2010 Feb;38(2):438-44. doi: 10.1097/CCM.0b013e3181b9eb3b. PMID 19789449
- [Background] Bagshaw SM, Lapinsky S, Dial S, Arabi Y, Dodek P, Wood G, Ellis P, Guzman J, Marshall J, Parrillo JE, Skrobik Y, Kumar A; Cooperative Antimicrobial Therapy of Septic Shock (CATSS) Database Research Group. Acute kidney injury in septic shock: clinical outcomes and impact of duration of hypotension prior to initiation of antimicrobial therapy. Intensive Care Med. 2009 May;35(5):871-81. doi: 10.1007/s00134-008-1367-2. Epub 2008 Dec 9. PMID 19066848
- [Background] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034
- [Background] Hernandez G, Ospina-Tascon GA, Damiani LP, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Granda-Luna V, Cavalcanti AB, Bakker J; The ANDROMEDA SHOCK Investigators and the Latin America Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon G, Petri Damiani L, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Cavalcanti AB, Bakker J, Hernandez G, Alegria L, Ferri G, Rodriguez N, Holger P, Soto N, Pozo M, Bakker J, Cook D, Vincent JL, Rhodes A, Kavanagh BP, Dellinger P, Rietdijk W, Carpio D, Pavez N, Henriquez E, Bravo S, Valenzuela ED, Vera M, Dreyse J, Oviedo V, Cid MA, Larroulet M, Petruska E, Sarabia C, Gallardo D, Sanchez JE, Gonzalez H, Arancibia JM, Munoz A, Ramirez G, Aravena F, Aquevedo A, Zambrano F, Bozinovic M, Valle F, Ramirez M, Rossel V, Munoz P, Ceballos C, Esveile C, Carmona C, Candia E, Mendoza D, Sanchez A, Ponce D, Ponce D, Lastra J, Nahuelpan B, Fasce F, Luengo C, Medel N, Cortes C, Campassi L, Rubatto P, Horna N, Furche M, Pendino JC, Bettini L, Lovesio C, Gonzalez MC, Rodruguez J, Canales H, Caminos F, Galletti C, Minoldo E, Aramburu MJ, Olmos D, Nin N, Tenzi J, Quiroga C, Lacuesta P, Gaudin A, Pais R, Silvestre A, Olivera G, Rieppi G, Berrutti D, Ochoa M, Cobos P, Vintimilla F, Ramirez V, Tobar M, Garcia F, Picoita F, Remache N, Granda V, Paredes F, Barzallo E, Garces P, Guerrero F, Salazar S, Torres G, Tana C, Calahorrano J, Solis F, Torres P, Herrera L, Ornes A, Perez V, Delgado G, Lopez A, Espinosa E, Moreira J, Salcedo B, Villacres I, Suing J, Lopez M, Gomez L, Toctaquiza G, Cadena Zapata M, Orazabal MA, Pardo Espejo R, Jimenez J, Calderon A, Paredes G, Barberan JL, Moya T, Atehortua H, Sabogal R, Ortiz G, Lara A, Sanchez F, Hernan Portilla A, Davila H, Mora JA, Calderon LE, Alvarez I, Escobar E, Bejarano A, Bustamante LA, Aldana JL. Effect of a Resuscitation Strategy Targeting Peripheral Perfusion Status vs Serum Lactate Levels on 28-Day Mortality Among Patients With Septic Shock: The ANDROMEDA-SHOCK Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):654-664. doi: 10.1001/jama.2019.0071. PMID 30772908
- [Background] Asfar P, Meziani F, Hamel JF, Grelon F, Megarbane B, Anguel N, Mira JP, Dequin PF, Gergaud S, Weiss N, Legay F, Le Tulzo Y, Conrad M, Robert R, Gonzalez F, Guitton C, Tamion F, Tonnelier JM, Guezennec P, Van Der Linden T, Vieillard-Baron A, Mariotte E, Pradel G, Lesieur O, Ricard JD, Herve F, du Cheyron D, Guerin C, Mercat A, Teboul JL, Radermacher P; SEPSISPAM Investigators. High versus low blood-pressure target in patients with septic shock. N Engl J Med. 2014 Apr 24;370(17):1583-93. doi: 10.1056/NEJMoa1312173. Epub 2014 Mar 18. PMID 24635770
- [Background] Lamontagne F, Richards-Belle A, Thomas K, Harrison DA, Sadique MZ, Grieve RD, Camsooksai J, Darnell R, Gordon AC, Henry D, Hudson N, Mason AJ, Saull M, Whitman C, Young JD, Rowan KM, Mouncey PR; 65 trial investigators. Effect of Reduced Exposure to Vasopressors on 90-Day Mortality in Older Critically Ill Patients With Vasodilatory Hypotension: A Randomized Clinical Trial. JAMA. 2020 Mar 10;323(10):938-949. doi: 10.1001/jama.2020.0930. PMID 32049269
- [Background] Lat I, Coopersmith CM, De Backer D, Coopersmith CM; Research Committee of the Surviving Sepsis Campaign. The surviving sepsis campaign: fluid resuscitation and vasopressor therapy research priorities in adult patients. Intensive Care Med Exp. 2021 Mar 1;9(1):10. doi: 10.1186/s40635-021-00369-9. PMID 33644843
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Saugel B, Vincent JL, Wagner JY. Personalized hemodynamic management. Curr Opin Crit Care. 2017 Aug;23(4):334-341. doi: 10.1097/MCC.0000000000000422. PMID 28562384
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Gleeson PJ, Crippa IA, Mongkolpun W, Cavicchi FZ, Van Meerhaeghe T, Brimioulle S, Taccone FS, Vincent JL, Creteur J. Renin as a Marker of Tissue-Perfusion and Prognosis in Critically Ill Patients. Crit Care Med. 2019 Feb;47(2):152-158. doi: 10.1097/CCM.0000000000003544. PMID 30653055
- [Background] Jeyaraju M, McCurdy MT, Levine AR, Devarajan P, Mazzeffi MA, Mullins KE, Reif M, Yim DN, Parrino C, Lankford AS, Chow JH. Renin Kinetics Are Superior to Lactate Kinetics for Predicting In-Hospital Mortality in Hypotensive Critically Ill Patients. Crit Care Med. 2022 Jan 1;50(1):50-60. doi: 10.1097/CCM.0000000000005143. PMID 34166293
- [Background] Kullmar M, Saadat-Gilani K, Weiss R, Massoth C, Lagan A, Cortes MN, Gerss J, Chawla LS, Fliser D, Meersch M, Zarbock A. Kinetic Changes of Plasma Renin Concentrations Predict Acute Kidney Injury in Cardiac Surgery Patients. Am J Respir Crit Care Med. 2021 May 1;203(9):1119-1126. doi: 10.1164/rccm.202005-2050OC. PMID 33320784
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Background] Semler MW, Rice TW, Shaw AD, Siew ED, Self WH, Kumar AB, Byrne DW, Ehrenfeld JM, Wanderer JP. Identification of Major Adverse Kidney Events Within the Electronic Health Record. J Med Syst. 2016 Jul;40(7):167. doi: 10.1007/s10916-016-0528-z. Epub 2016 May 27. PMID 27234478
- [Background] Kotani Y, Landoni G, Belletti A, Khanna AK. Response to: norepinephrine formulation for equivalent vasopressive score. Crit Care. 2023 Mar 28;27(1):125. doi: 10.1186/s13054-023-04404-x. No abstract available. PMID 36978126
- [Background] Kotani Y, Belletti A, D'Andria Ursoleo J, Salvati S, Landoni G. Norepinephrine Dose Should Be Reported as Base Equivalence in Clinical Research Manuscripts. J Cardiothorac Vasc Anesth. 2023 Sep;37(9):1523-1524. doi: 10.1053/j.jvca.2023.05.013. Epub 2023 May 11. No abstract available. PMID 37291003